CLINICAL TRIAL: NCT03594071
Title: Safety and Performance of Q-Fix™ All-Suture Anchor System
Brief Title: S&P of Q-Fix™ All-Suture Anchor System
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-5010-11
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Bankart Lesion; Acetabular Labrum Tear; SLAP Lesion; Acromioclavicular Sprain; Capsular Shift/Capsulolabral Reconstruction; Deltoid Repair; Rotator Cuff Repair; Bicep Tendinitis; Extra-capsular Repair; Medial Collateral Ligament; Lateal Collateral Ligament; Posterior Oblique Ligament; IBT; Vastus Medialis; Obliquus Advancement; Joint Capsule Closure
MeSH Terms: conditions — Bankart Lesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: The Q-Fix™ All-Suture Anchor — Observational, post-market, clinical follow-up study

SUMMARY:
Post-market clinical follow-up needed to address existing clinical data and gaps on the existing Q-Fix™ device and meet existing MDD/MEDDEV requirements

ELIGIBILITY:
Inclusion Criteria:

* Subject has undergone arthroscopic or open soft tissue repair with Q-Fix™ All-Suture Anchor System
* Subject was ≥ 13 of age at time of surgery

Exclusion Criteria:

* Subject is ≤ 6 months post-operative
* Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 12 months post-operative.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: US sites
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Langone, Study Chair — GBR - T. J. Smith and Nephew Limited
Locations (5):
- United States (5):
  - The Orthopaedic Center- Center for Advanced Orthopaedics, Washington D.C., District of Columbia
  - Northshore University Health System, Chicago, Illinois
  - Tulane University Medical Center /Tulane Institute of Sport Medicine, New Orleans, Louisiana
  - Oklahoma Sports and Orthopedics Institute, Oklahoma City, Oklahoma
  - Palmetto Health USC Orthopedic Center, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No
* Study Protocol
  * Clinical Study Report (CSR)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 294 subjects at 5 investigational sites in the United States. This included a total of 309 joints: 134 hips, 118 shoulders, and 57 knees.
Units Other Than Participants: joints
Groups:
- Safety Population: All subjects enrolled into the study
Period: Overall Study
Arm/Group | Safety Population
Started | 294; 309 joints
Completed | 289; 304 joints
Not Completed | 5; 5 joints
Not completed — Re-operation | 3
Not completed — Missed visit | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 294
Number analyzed (joints) | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.10 (16.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 147
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 228
  Asian | 4
  Black or African American | 29
  American Indian or Alaska Native | 4
  Other | 7
  Unknown | 22
Region of Enrollment [Number; unit: participants]
  United States | 294
Height [Mean (Standard Deviation); unit: cm] — Population: Includes all data available for this particular measure (retrospective data)
  cm
    number analyzed (Participants) | 289
    (all) | 171.19 (11.449)
Weight [Mean (Standard Deviation); unit: pounds (lb)] — Population: Includes all data available for this particular measure (retrospective data)
  pounds (lb)
    number analyzed (Participants) | 288
    (all) | 177.33 (46.045)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Includes all data available for this particular measure (retrospective data)
  kg/m^2
    number analyzed (Participants) | 287
    (all) | 27.39 (7.060)
Ethnicity [Count of Participants; unit: Participants] — Population: Includes all data available for this particular measure (retrospective data)
  Participants
    number analyzed (Participants) | 257
    Hispanic/Latino | 15
    Not Hispanic/Latino | 242

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success Rate, Defined as Participant Joints Without Reintervention at 6 Months Post-operative, as Assessed by the Surgeon
Description: All individuals for whom the outcome of re-intervention is known at 6 months
Time Frame: 6 months
Population: Per Safety Population, this includes all participants who enrolled in the study who had previously undergone arthroscopic repair using the Q-Fix™ All-Suture Anchor System (i.e. participants that provided retrospective data at the time frame indicated)
Measure: Count of Units; unit: joints
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 294
Number analyzed (joints) | 309
joints | 306

2. Secondary Outcome: Clinical Success Rate, Defined as Participant Joints Without Reintervention at 12 Months Post-operative, as Assessed by the Surgeon
Description: All individuals for whom the outcome of re-intervention is known at 12 months
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Units; unit: joints
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 109
Number analyzed (joints) | 122
joints | 118

3. Secondary Outcome: Hip Visual Analog Scale (VAS) - Pain
Description: VAS scores as reported by the site were converted if required such that all data was reported on a scale of 0-100 (e.g. if the scale was 0-10, then the value was multiplied by 10). Note that VAS scores should be interpreted with caution as use of pain medications may affect the results. A higher score indicates more pain.
Time Frame: Screening, 6 months, and 12 months
Population: Per Safety Population, this includes all participants who enroll in the study who had previously undergone arthroscopic repair using the Q-Fix™ All-Suture Anchor System i.e. subjects who only provide retrospective data.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 113
Number analyzed (joints) | 119
score on a scale
  Hip: Screening | 51.0 (21.7)
  Hip: 6 months: number analyzed (Participants) | 69
  Hip: 6 months: number analyzed (joints) | 71
  Hip: 6 months | 24.4 (20.7)
  Hip: 12 months: number analyzed (Participants) | 32
  Hip: 12 months: number analyzed (joints) | 32
  Hip: 12 months | 16.3 (18.3)

4. Secondary Outcome: Knee Visual Analog Scale (VAS) - Pain
Description: as for outcome 3
Time Frame: Screening, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 8
Number analyzed (joints) | 8
score on a scale
  Knee: Screening | 51.3 (25.3)
  Knee: 6 months: number analyzed (Participants) | 3
  Knee: 6 months: number analyzed (joints) | 3
  Knee: 6 months | 10.0 (17.3)
  Knee: 12 months: number analyzed (Participants) | 3
  Knee: 12 months: number analyzed (joints) | 3
  Knee: 12 months | 23.3 (40.4)

5. Secondary Outcome: Shoulder Visual Analog Scale (VAS) - Pain
Description: as for outcome 3
Time Frame: Screening, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 51
Number analyzed (joints) | 51
score on a scale
  Shoulder: Screening | 53.3 (26.4)
  Shoulder: 6 months: number analyzed (Participants) | 37
  Shoulder: 6 months: number analyzed (joints) | 37
  Shoulder: 6 months | 28.8 (25.4)
  Shoulder: 12 months: number analyzed (Participants) | 9
  Shoulder: 12 months: number analyzed (joints) | 9
  Shoulder: 12 months | 35.6 (27.4)

6. Secondary Outcome: Hip Range of Motion (ROM)
Description: Full Range of Motion (ROM) defined as full functional arc in hip by the physician.
Time Frame: Screening, 6 months, and 12 months
Population: as for outcome 1
Measure: Count of Units; unit: joints
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 120
Number analyzed (joints) | 134
joints
  Hip: Screening - has full functional arc: number analyzed (Participants) | 119
  Hip: Screening - has full functional arc: Yes | 37
  Hip: Screening - has full functional arc: No | 90
  Hip: Screening - has full functional arc: Missing | 7
  Hip: 6 months- has full functional arc: number analyzed (joints) | 133
  Hip: 6 months- has full functional arc: Yes | 45
  Hip: 6 months- has full functional arc: No | 81
  Hip: 6 months- has full functional arc: Missing | 7
  Hip: 12 months- has full functional arc: number analyzed (Participants) | 70
  Hip: 12 months- has full functional arc: number analyzed (joints) | 78
  Hip: 12 months- has full functional arc: Yes | 32
  Hip: 12 months- has full functional arc: No | 42
  Hip: 12 months- has full functional arc: Missing | 4

7. Secondary Outcome: Knee Range of Motion (ROM)
Description: Full Range of Motion (ROM) defined as full functional arc in knee by the physician
Time Frame: Screening, 6 months, and 12 months
Population: as for outcome 1
Measure: Count of Units; unit: joints
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 47
Number analyzed (joints) | 57
joints
  Knee: Screening - has full functional arc: number analyzed (Participants) | 39
  Knee: Screening - has full functional arc: Yes | 28
  Knee: Screening - has full functional arc: No | 14
  Knee: Screening - has full functional arc: Missing | 15
  Knee: 6 months- has full functional arc: number analyzed (joints) | 56
  Knee: 6 months- has full functional arc: Yes | 24
  Knee: 6 months- has full functional arc: No | 25
  Knee: 6 months- has full functional arc: Missing | 7
  Knee: 12 months- has full functional arc: number analyzed (Participants) | 13
  Knee: 12 months- has full functional arc: number analyzed (joints) | 14
  Knee: 12 months- has full functional arc: Yes | 7
  Knee: 12 months- has full functional arc: No | 6
  Knee: 12 months- has full functional arc: Missing | 1

8. Secondary Outcome: Shoulder Range of Motion (ROM)
Description: Full Range of Motion (ROM) defined as full functional arc in shoulder by the physician.
Time Frame: Screening, 6 months, and 12 months
Population: as for outcome 1
Measure: Count of Units; unit: joints
Units Other Than Participants: joints
Arm/Group | Safety Population
Number analyzed (Participants) | 112
Number analyzed (joints) | 118
joints
  Shoulder: Screening - has full functional arc: Yes | 14
  Shoulder: Screening - has full functional arc: No | 100
  Shoulder: Screening - has full functional arc: Missing | 4
  Shoulder: 6 months- has full functional arc: number analyzed (joints) | 115
  Shoulder: 6 months- has full functional arc: Yes | 24
  Shoulder: 6 months- has full functional arc: No | 90
  Shoulder: 6 months- has full functional arc: Missing | 1
  Shoulder: 12 months- has full functional arc: number analyzed (Participants) | 24
  Shoulder: 12 months- has full functional arc: number analyzed (joints) | 27
  Shoulder: 12 months- has full functional arc: Yes | 8
  Shoulder: 12 months- has full functional arc: No | 16
  Shoulder: 12 months- has full functional arc: Missing | 3

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/294
Serious Adverse Events (participants affected / at risk) | 22/294
Other Adverse Events (participants affected / at risk) | 81/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=294)
Abcess of shoulder (Infections and infestations) | 1 (1) — Unrelated to device
Adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Related to device
Biceps tear/tendon rupture (Injury, poisoning and procedural complications) | 2 (2) — Unrelated to device
Biceps tear/tendon rupture (Injury, poisoning and procedural complications) | 2 (2) — Possibly related to device
Biceps tear/tendon rupture (Injury, poisoning and procedural complications) | 1 (1) — Related to device
Bone fracture (Injury, poisoning and procedural complications) | 2 (2) — Unrelated to device
Graves disease (General disorders) | 1 (1) — Unrelated to device
Hip pain (General disorders) | 1 (1) — Related to device
Hip pain (General disorders) | 1 (1) — Unrelated to device
Incomplete healing (General disorders) | 1 (1) — Unrelated to device
Knee Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 2 (3) — Unrelated to device
Labral tear (Injury, poisoning and procedural complications) | 1 (1) — Unrelated to device
Recurrent rotator cuff tear (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Unrelated to device
Removal of screw (Congenital, familial and genetic disorders) | 1 (1) — Unrelated to device
Rotator cuff and slap lesion repair (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated to device
Shoulder Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Spinal cyst (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Suicidal ideation (Psychiatric disorders) | 1 (1) — Unrelated to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=294)
Abdominal pain (General disorders) | 1 (1) — Unrelated to device
Adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated to device
Arm pain (General disorders) | 1 (1) — Unrelated to device
Back pain (General disorders) | 2 (2) — Unrelated to device
Clicking/popping sensation (Musculoskeletal and connective tissue disorders) | 7 (7) — Unrelated to device
Clicking/popping sensation (Musculoskeletal and connective tissue disorders) | 4 (4) — Possibly related to device
Constipation (Gastrointestinal disorders) | 1 (1) — Unrelated to device
Discoloration of foot (General disorders) | 1 (1) — Unrelated to device
Erythema/rash (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated to device
Groin pain (General disorders) | 3 (3) — Unrelated to device
Groin pain (General disorders) | 1 (1) — Possibly related to device
Groin stiffness/tightness (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated to device
Hematuria (Renal and urinary disorders) | 1 (1) — Unrelated to device
Hip pain (General disorders) | 19 (23) — Unrelated to device
Hip pain (General disorders) | 2 (2) — Possibly related to device
Hip stiffness/tightness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Implant pulled out of bone (Injury, poisoning and procedural complications) | 1 (1) — Related to device
Inflammation (General disorders) | 2 (3) — Unrelated to device
Injury (Injury, poisoning and procedural complications) | 8 (10) — Unrelated to device
Knee pain (General disorders) | 2 (2) — Unrelated to device
Leg pain (General disorders) | 6 (6) — Unrelated to device
Leg pain (General disorders) | 1 (1) — Possibly related to device
Lumbar facet arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Lymphedema (General disorders) | 1 (1) — Unrelated to device
Muscle strain (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated to device
Numbness/weakness (General disorders) | 8 (8) — Unrelated to device
Pain (General disorders) | 4 (5) — Unrelated to device
Pain (General disorders) | 1 (1) — Possibly related to device
Patellar malalignment (Nervous system disorders) | 1 (1) — Unrelated to device
Recurrent shoulder instability (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated to device
Shoulder pain (General disorders) | 5 (6) — Unrelated to device
Shoulder pain (General disorders) | 1 (1) — Possibly related to device
Shoulder subluxation (Injury, poisoning and procedural complications) | 1 (1) — Unrelated to device
Snapping Iliopsoas Tendon (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated to device
Stiffness/tightness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to device
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Unrelated to device
Withdrawal symptoms (General disorders) | 1 (1) — Unrelated to device
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) — Unrelated to device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03594071/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT03594071/SAP_001.pdf